CLINICAL TRIAL: NCT05459311
Title: Investigating Radiation-Induced Injury to Airways and Pulmonary Vasculature in Lung Stereotactic Ablative Body Radiotherapy (SAbR)
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU-062016-073
Record Dates: First submitted 2022-06-10; First posted 2022-07-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer; Thoracic Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will conduct a prospective clinical study involving up to 40 non-Small Cell Lung Cancer (nSCLC) patients to determine dose thresholds for central and peripheral BSS elements. All imaging will be performed under motion control (e.g., with or without abdominal compression) defined as breathing with a resultant motion ≤5mm by fluoroscopy.

In this study, a high-resolution breath-hold CT scan (BHCT) will be acquired from each patient immediately before or after the 4DCT scan.

A follow-up high resolution BHCT (also under motion control) will be acquired from each patient 8-12 months post-SabR, and BSS elements will be segmented in LungPointRT. A radiation oncologist will compare the pre- and post-SabR contours to determine segmental collapse.

DETAILED DESCRIPTION:
We will conduct a prospective clinical study involving up to 40 non-Small Cell Lung Cancer (nSCLC) patients to determine dose thresholds for central and peripheral BSS elements. The workflow is illustrated in Fig. 4. all imaging will be performed under motion control (e.g., with or without abdominal compression) defined as breathing with a resultant motion [LessThanorequalTo]5mm by fluoroscopy. Before 4DCT simulation, fluoroscopy using a stand-alone system is used to assess motion under free-breathing conditions. For those with inherent motion [LessThanorequalTo]5mm, no motion manipulation is required (ie, motion is controlled). For those with [Greater Than]5mm motion, it is customary to use progressively tighter abdominal compression applied via commercially available device or a pneumatic belt, until respiration-induced tumor motion, as seen under fluoroscopy, is [LessThanorequalTo] 5mm. Subsequently, a 4DCT scan is acquired with motion control.

in this study, a high-resolution breath-hold CT scan (BHCT) will be acquired from each patient immediately before or after the 4DCT scan. using LungPoint, a virtual bronchoscopy software, individual BSS will be auto-segmented from the BHCT, labeled based on a nomenclature described by netter and exported as Digital imaging and Communications in Medicine radiation Therapy (DiCoMRT) objects to the planning system. The BHCT will be deformably registered to each phase of the 4DCT to create ten high-resolution CT volumes corresponding to ten respiratory phases. acquiring both, the BHCT and the 4DCT, under motion control will ensure that the anatomy is consistently deformed so as to minimize image registration errors. The automatically deformed contours, especially for smaller BSS elements, will be manually verified by a radiation oncologist, and corrected if necessary. a high-resolution maximum intensity projection (MiP) image will be created from the deformed BHCT volumes so as to encompass the extent of respiration-induced motion for each structure in the lung. The high spatial resolution of the MiP will ensure that respiratory motion of smaller, more peripheral BSS segments is captured accurately. The dose to BSS elements from the clinical SabR plan (created without considering BSS) will be computed from the hi-res MiP using the acuros dose calculation algorithm. This algorithm accurately accounts for dose to small structures and tissue inhomogeneities, and has been extensively validated for lung radiotherapy.

a follow-up high resolution BHCT (also under motion control) will be acquired from each patient 8-12 months post-SabR, and BSS elements will be segmented in LungPointRT. a radiation oncologist will compare the pre- and post-SabR contours to determine segmental collapse. univariate and multivariate stepwise generalized estimating equation (Gee) analyses will be conducted to identify significant factors contributing to BSS collapse, accounting for intra-patient correlation within each nSCLC patient. The insights obtained from these analyses will be used to formulate dose-thresholds for BSS segments. For each segment, we will compute the probability of segmental collapse as a function of dose, Cs(D) and also assign a weight [and] #955;s. This weight will be based on the findings of aim 2 and will be proportional to the functional lung volume [Quote]served[Quote] by that segment. This weighting scheme will ensure that the dose-thresholds (DT) are set more conservatively, i.e., with relatively lower Cs(DT) for the more critical BSS segments and vice versa.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary or metastatic lesions in the lung, to be treated with definitive proton or photon radiotherapy. There is no limitation on the number of radiotherapy fractions, or the location/number of lesions for this study
2. Age ≥ 18 years. No gender or ethnic restrictions.
3. ECOG performance status ≤ 3
4. Ability to hold breath for ~20 seconds
5. Ability to understand and the willingness to sign a written informed consent.
6. Any types and amounts of prior therapy will be allowed for this study.
7. All men, as well as women of child-bearing potential must agree to use adequate contraception (surgical sterilization [hysterectomy or vasectomy], approved hormonal contraceptives [birth control pills, patch or ring, Depo-Provera, Implanon] or barrier method such as condom or diaphragm with spermicide or an intrauterine device) from consent until the end of study scans. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   * A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

     * Has not undergone a hysterectomy or bilateral oophorectomy; or
     * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Children (age <18 years).
2. Women who are pregnant, nursing, or trying to get pregnant
3. ECOG performance status > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Lung/Thoracic malignancies who consent to recieving Radiation treatment at the University of Texas Medical Center, will be offered this protocol design.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
The association between radiation-induced collapse of Branching Serial Structures (BSS) elements and localized change in pulmonary function. | 24 months
  Evaluating the association between radiation-induced collapse of Branching Serial Structures (BSS) elements, characterized by segmental collapse, and localized change in pulmonary function. a map of collapsed and open BSS elements will be generated from the contoured BSS trees in the pre- and post-SAbR BHCT scans to determine the impact of radiation-induced collapse of BSS elements and localized changes to pulmonary function.
The radiosensitivity of peripheral Branching Serial Structures (BSS) segments. | 24 months
  Evaluating the radiosensitivity of peripheral BSS segments in terms of dose dependent probability of collapse through Generalized Estimating Equation (GEE).

SECONDARY OUTCOMES:
Create intensity modulated radiotherapy treatment plans | 24 months
  To create intensity modulated radiotherapy treatment plans that incorporate radiation dose thresholds for BSS elements while achieving other clinical objectives (prescription dose to planning target volume, dose limits to other organs at risk).

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Cancer Center, Dallas, Texas, United States